CLINICAL TRIAL: NCT07375940
Title: Clinical, Biochemical and Epigenetic Profile of Pediatric Behçet Disease: Similarities and Differences From Adult Patients and Looking for Potential Biomarkers.
Brief Title: Clinical, Biochemical and Epigenetic Profile of Pediatric Behçet Disease
Acronym: PED-BD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Gabriele Simonini, MD, Meyer Children's Hospital IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PED-BD
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Behcet Disease and Vascular Involvement
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pediatric Behçet Disease Patients (Other): Pediatric patients (<18 years) with a diagnosis of Behçet disease. Blood samples collected during routine clinical visits will be analyzed for research purposes, including cytokine profiling, circulating microRNA analysis, DNA methylation profiling, and genetic sequencing. These analyses are not used for clinical decision-making.
  Interventions: Diagnostic Test: Biomarker analysis of blood samples
- Adult Behçet Disease Patients (Experimental): Adult patients (≥18 years) with a diagnosis of Behçet disease. Blood samples collected during routine clinical visits will be analyzed for research purposes, including cytokine profiling, circulating microRNA analysis, DNA methylation profiling, and genetic sequencing. These analyses are not used for clinical decision-making
  Interventions: Diagnostic Test: Biomarker analysis of blood samples
- Healthy Pediatric Controls (Experimental): Healthy pediatric subjects (<18 years) undergoing routine blood testing for non-inflammatory conditions. Blood samples will be analyzed for research purposes, including circulating microRNA analysis and DNA methylation profiling, and used as reference controls for comparative analyses.
  Interventions: Diagnostic Test: Biomarker analysis of blood samples

INTERVENTIONS:
Diagnostic Test: Biomarker analysis of blood samples — Research laboratory analyses will be performed on blood samples collected during routine clinical care.
  For pediatric Behçet disease patients, analyses include cytokine profiling (IL-6, IL-10, IL-17, TNF-α), circulating microRNA profiling, DNA methylation profiling, and targeted genetic sequencing for genes associated with monogenic Behçet-like phenotypes.
  Arms: Healthy Pediatric Controls
Diagnostic Test: Biomarker analysis of blood samples — Research laboratory analyses will be performed on blood samples collected during routine clinical care.
  For Adult Behçet disease patients, analyses include cytokine profiling (IL-6, IL-10, IL-17, TNF-α), circulating microRNA profiling, DNA methylation profiling, and targeted genetic sequencing for genes associated with monogenic Behçet-like phenotypes.
  Arms: Adult Behçet Disease Patients
Diagnostic Test: Biomarker analysis of blood samples — Research laboratory analyses will be performed on blood samples collected during routine clinical care.
  For healthy pediatric controls, analyses are limited to circulating microRNA profiling and DNA methylation profiling only; no genetic testing/DNA sequencing will be performed in this group.
  Arms: Pediatric Behçet Disease Patients

SUMMARY:
Behçet disease (BD) is a chronic multisystem inflammatory disorder with a relapsing-remitting course. Pediatric-onset BD is rare and characterized by marked clinical heterogeneity, frequent incomplete presentation at disease onset, and limited availability of pediatric-specific outcome measures and biomarkers.

This prospective multicenter study aims to comprehensively characterize the clinical, biochemical, genetic, and epigenetic profiles of pediatric patients with Behçet disease and to compare them with adult BD patients and healthy pediatric controls.

The study focuses on the identification of disease-associated cytokine patterns, circulating microRNA profiles, DNA methylation signatures, and genetic variants associated with monogenic autoinflammatory diseases presenting with a Behçet-like phenotype.

By integrating clinical data with multi-omic analyses, this study seeks to identify biologically and clinically meaningful patient subgroups, improve disease stratification, and explore potential biomarkers of disease activity and remission in pediatric Behçet disease.

DETAILED DESCRIPTION:
Behçet disease is a chronic inflammatory disorder involving mucocutaneous, ocular, vascular, neurological, gastrointestinal, and musculoskeletal systems. Although the clinical manifestations of pediatric BD are largely similar to those observed in adults, pediatric cases show greater heterogeneity, higher familial aggregation, and frequent diagnostic uncertainty, particularly at early disease stages.

The etiopathogenesis of BD remains incompletely understood and is thought to involve a complex interaction between genetic predisposition, immune dysregulation, environmental triggers, and epigenetic mechanisms. Increased levels of pro-inflammatory cytokines, including interleukin (IL)-6, IL-17, and tumor necrosis factor alpha (TNF-α), as well as altered circulating microRNA and DNA methylation profiles, have been reported in adult BD patients, but data in pediatric populations are scarce.

This prospective, multicenter, case-control study will enroll pediatric and adult patients with Behçet disease and healthy pediatric controls. Clinical data will be collected longitudinally, and biological samples will be obtained during routine blood draws at predefined disease stages, including diagnosis, sustained remission, and disease flare.

The study will evaluate circulating cytokine levels, genome-wide DNA methylation profiles, circulating microRNAs, and genetic variants associated with monogenic autoinflammatory diseases that can mimic BD. Pediatric healthy controls will provide reference epigenetic and microRNA profiles for comparative analyses.

Through integrated clinical and molecular analyses, this study aims to identify disease-associated molecular signatures, characterize patient subgroups, and improve understanding of pediatric Behçet disease pathogenesis, potentially supporting future development of personalized diagnostic and therapeutic strategies.

ELIGIBILITY:
Cases Inclusion Criteria :

* BD diagnosis according to at least one of the three sets of classification criteria [International Criteria for Behçet's Disease (ICBD), International Study Group (ISG) and Pediatric Behçet's disease criteria PEDBD)];
* Age 6 months to 70 years old.
* Written informed consent from appropriate legal representative(s), and assent from patients who have not reached the age of consent.

Cases Exclusion Criteria:

* Patients who do not meet the BD criteria OR
* Patients for whom an alternative diagnosis was not investigated and/or excluded OR
* Absence of a written informed consent.

Healthy pediatric controls:

* Patients evaluated at the Meyer Children's Hospital IRCCS Rheumatology Outpatient Clinic who are scheduled to undergo routine hematochemical tests, not for suspected inflammatory or autoimmune conditions.
* Age < 18 years, matched 1:1 by age and sex with the pediatric Behçet disease (BD) cohort.
* Absence of recent or ongoing inflammatory conditions, verified through structured medical history and physical examination.
* No clinical signs suggestive of chronic autoinflammatory or autoimmune diseases at physical examination .
* No recent prolonged use (more than 7 consecutive days within the past 4 weeks) of anti-inflammatory, glucocorticoids, immunomodulatory, therapies or antibiotics.
* Written informed consent from the legal guardian(s) and assent from minors when appropriate.

Healthy Controls Exclusion Criteria

* Diagnosis of acute or chronic inflammatory, autoimmune, or autoinflammatory conditions after the collection of structured medical history and physical examination
* Current or recent prolonged use (more than 7 consecutive days within the past 4 weeks) of anti-inflammatory drugs, gluccocorticoids, immunomodulatory agents, or antibiotics.
* Routine blood tests not performed during the visit.
* Absence of written informed consent.

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2036-01 (Estimated); Study Completion 2036-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative biomarker profiles in Behçet disease | Up to 24 months
  Quantitative measurement of circulating biomarker levels in blood samples, including serum cytokine concentrations (IL-6, IL-10, IL-17, TNF-α), circulating microRNA expression levels, DNA methylation beta values at genome-wide CpG sites, and presence or absence of pathogenic genetic variants associated with monogenic Behçet-like diseases.
  Biomarker measurements will be obtained in pediatric and adult patients with Behçet disease and, where applicable, compared with healthy pediatric controls to evaluate differences across disease status and age groups.

SECONDARY OUTCOMES:
Circulating microRNA expression levels | Up to 24 months
  Quantitative assessment of circulating microRNA expression levels in plasma samples obtained from pediatric and adult patients with Behçet disease and healthy pediatric controls, measured using microarray-based profiling and validation assays.
Genome-wide DNA methylation beta values | Up to 24 months
  Quantitative measurement of genome-wide DNA methylation beta values at CpG sites in genomic DNA extracted from blood samples collected from pediatric and adult patients with Behçet disease and healthy pediatric controls.
Serum cytokine concentrations in Behçet disease | Up to 24 months
  Quantitative measurement of serum cytokine concentrations, including interleukin-6 (IL-6), interleukin-10 (IL-10), interleukin-17 (IL-17), and tumor necrosis factor alpha (TNF-α), measured in blood samples collected from pediatric and adult patients with Behçet disease during diagnosis, disease flare, and sustained remission.
Presence of pathogenic genetic variants associated with Behçet-like phenotypes | Baseline
  Detection and quantification of the presence or absence of pathogenic or likely pathogenic genetic variants in genes associated with monogenic autoinflammatory diseases presenting with a Behçet-like phenotype, assessed through targeted next-generation sequencing in pediatric and adult patients with Behçet disease.

CONTACTS AND LOCATIONS:
Locations (2):
- Aou Meyer IRCSS, Florence, Florence, Italy
- Alder Hey Children's Hospital,, Liverpool, Liverpool, United Kingdom